CLINICAL TRIAL: NCT04182412
Title: Minimally Invasive Abdominal Wall Reconstruction in Symptomatic Rectus Diastasis
Brief Title: Abdominal Rectus Diastasis (ARD) Reconstruction
Acronym: ARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Thorell, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-01959
Record Dates: First submitted 2019-11-07; First posted 2019-12-02 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Rectus Diastasis
Keywords: Laparoscopy; mesh reinforcement; abdominal stability

STUDY DESIGN:
Intervention Model Description: two different laparoscopic to one of techniques for abdominal wall reconstruction: narrowing of linea alba with continuous suture, with and without mesh
Who Masked: Participant, Investigator
Masking Description: The randomization process will be initiated after general anesthesia is induced and the group affiliation will be determined by opening of a sealed envelope specifying the group assignment. The information of group allocation is stored in a closed envelope kept in a locked archive until the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture (Active Comparator): laparoscopic narrowing of linea alba with continuous suture
  Interventions: Procedure: ARD
- suture and mesh (Active Comparator): narrowing of linea alba with continuous suture and mesh
  Interventions: Procedure: ARD

INTERVENTIONS:
Procedure: ARD — surgical reconstruction with laparoscopic technique

SUMMARY:
The aim of this study is to investigate whether abdominal wall reconstruction through laparoscopic surgery can be recommended as a safe treatment alternative for patients with symptomatic rectus diastasis, and if this type of treatment leads to improved quality of life, trunk stability and reduced pain.

DETAILED DESCRIPTION:
Investigate whether surgical reconstruction with laparoscopic technique can lead to improved quality of Life, trunk stability and reduced pain in patients with symptomatic rectus diastasis. The study will also compare two different laparoscopic surgery methods for abdominal wall reconstruction: narrowing of linea alba with continuous suture with or without mesh.

ELIGIBILITY:
Inclusion Criteria:

* Rectus diastasis ≥3 cm
* BMI =<28 kg/m2
* non smoker
* abdominal instability,
* abdominal wall and/or lower back pain despite physical therapy / structured physical exercise for at least 6 months

Exclusion Criteria:

* BMI >28 kg/m2
* Smoking
* Ongoing immunosuppressive therapy
* Current pregnancy ≥16 weeks gestational age for the last 12 months
* Pregnant or women who wish to become pregnant
* Previously extensive abdominal wall surgery incl hernia surgery (NOT including sectio, appendectomy, small umbilical herniae)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence | 1 year
  computed tomography

SECONDARY OUTCOMES:
Visual Analog Pain Scale (VAS) | 1 year, 3 years
  Scale from 0 to 10, where 0 is no pain and 10 is the worst possible pain
Abdominal stability | 1 year, 3 years
  patient self-esteem by one question; do you feel that the instability of the abdominal wall has disappeared, yes/no/partially
SF-36 Quality of Life instrument | 1 year, 3 years
  The RAND-36 It is comprised of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. Higher scores mean a better outcome.
VHPQ is a questionnaire for the assessment of pre- and postoperative pain | 1 year, 3 years
  The questionnaire comprises 20 questions The first six questions concern the level and duration of pain. The next seven questionsrelate to the impact on daily activities. The final questions deal with patient satisfaction and how physically demanding the patients regard their occupation. Pain intensity in the VHPQ is assessed using a 7-step fixed-point rating scale with steps linked to pain behavior rather than numbers or verbal descriptors of pain. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Ersta Hospital, Stockholm, Region Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No